CLINICAL TRIAL: NCT06259292
Title: CHORUS: Comprehensive HHT (Hereditary Hemorrhagic Telangiectasia) Outcomes Registry of the United States
Brief Title: Comprehensive HHT Outcomes Registry of the United States (CHORUS)
Acronym: CHORUS
Status: Recruiting | Type: Observational
Sponsor: Cure HHT (Other)
Collaborators: Augusta University (Other); The Cleveland Clinic (Other); Mayo Clinic (Other); Massachusetts General Hospital (Other); Columbia University (Other); Oregon Health and Science University (Other); University of California, Los Angeles (Other); University of California, San Francisco (Other); University of Colorado, Denver (Other); University of North Carolina, Chapel Hill (Other); University of Pennsylvania (Other); University of Texas (Other); University of Utah (Other); Washington University School of Medicine (Other); Yale University (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: HHT001
Record Dates: First submitted 2024-01-22; First posted 2024-02-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Arteriovenous Malformations; Telangiectasia; Epistaxis; GastroIntestinal Bleeding; Cerebral Arteriovenous Malformations; Vascular Malformation
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Arteriovenous Malformations; Telangiectasis; Epistaxis; Gastrointestinal Hemorrhage; Intracranial Arteriovenous Malformations; Vascular Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HHT patients: Those diagnosed with HHT based on the Curacao diagnostic criteria or genetic testing

SUMMARY:
The Comprehensive HHT Outcomes Registry of the United States (CHORUS) is an observational registry of patients diagnosed with Hereditary Hemorrhagic Telangiectasia (HHT). The purpose of this study is to better understand HHT, the symptoms and complications it causes, and the impact the disease has on people's lives. The investigators will collect long-term information about the participant, allowing us to understand how the disease changes over time, and what factors can influence those changes. Ultimately, this should help improve treatments for the disease.

Another important goal of the study is to provide a way to contact people to participate in future clinical trials and other research. The registry will be a centralized resource for recruitment for clinical trials. People in the registry will not be obligated to join any of these additional studies, but if interested, can agree to be contacted if they may be eligible for a study.

Participants will:

* Be asked to provide permission to collect information from their medical records, including things like demographic information, diagnosis information, family history, test results, treatment information, symptoms, complications, lifestyle and other relevant medical information.
* Be asked study-related questions by phone or at a clinic visit.
* Be asked study-related questions every year after enrollment for up to 10 years or until the study ends. A member of the study team will communicate with participants by phone or at clinic visits to collect information regarding any changes to their health over the previous year/s including new test results, treatment information, symptoms, and complications from HHT.

DETAILED DESCRIPTION:
The Comprehensive HHT Outcomes Registry of the United States (CHORUS) is a research initiative led by the HHT Foundation International, Inc. ("Cure HHT"). The study focuses on Hereditary Hemorrhagic Telangiectasia (HHT), a rare genetic disorder characterized by the development of abnormal blood vessels in various organs of the body, including the brain, spine, lungs, liver, GI tract, skin, nasal mucosa, and oral cavity. The prevalence of HHT is estimated to be 1 in 5000, affecting children and adults. These abnormal blood vessels can lead to acute and chronic bleeding, stroke, heart failure, and death. Treatments are currently predominately limited to managing complications, while approximately 90% of adults have ongoing symptoms, despite the best surgical and medical therapies. With recent drug developments related to angiogenesis, there is hope for effective novel therapies.

A natural history registry for HHT has significant implications for improving the understanding and management of this rare genetic disorder. The purpose of this study is to better understand HHT, the symptoms and complications it causes ("outcomes"), and to understand how the disease impacts people's lives. The investigators hypothesize that a natural history registry for HHT will improve our understanding of the disease, lead to better management of patients, and ultimately, contribute to developing novel therapies to treat this disease.

The investigators will collaborate with multiple HHT Centers of Excellence across the U.S. to establish a comprehensive registry of HHT patients. The study aims to enroll approximately 10,000 HHT patients over a 10-year period. Longitudinal data will be collected both retrospectively and prospectively, with a focus on increasing the understanding of this rare disease, accelerating the development of new diagnostic and treatment options, and working collaboratively with clinicians who care for individuals with HHT to identify and address gaps in the system of care, especially those from underserved populations.

The study aims to serve as a centralized resource for future clinical trials and research in HHT. Data security and confidentiality are prioritized, and participants have the option to withdraw from the study at any time. The study is funded by the U.S. Department of Health Resources and Service Administration (HRSA) through a grant awarded to Cure HHT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HHT based on the Curacao diagnostic criteria or genetic testing.
* Able to provide informed consent or informed consent via a parent or legally authorized representative due to their age or medical condition.

Exclusion Criteria:

* Unable to provide informed consent or informed consent via a parent or legally authorized representative.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients evaluated and diagnosed with HHT in the U.S. will be eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2033-11 (Estimated); Study Completion 2033-11 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Baseline Data Collection using HHT Baseline Assessment Scale | 10 years
  Utilizing the "HHT Baseline Assessment Scale," this measure focuses on recruiting a diverse cohort of HHT patients across North America. Comprehensive baseline clinical, demographic, and lifestyle data will be collected and entered into CHORUS. The data, aggregated as mean change from baseline using the scale, will serve as a foundational resource for future clinical translational studies, addressing the urgent need for natural history data in HHT.
Prospective Longitudinal Clinical Outcomes Assessment using HHT Clinical Outcomes Scale | 10 years
  Utilizing the "HHT Clinical Outcomes Scale," this measure aims to prospectively and longitudinally assess the clinical outcomes of HHT patients. Determinants such as demographic factors, environmental influences, lifestyle choices, comorbidities, medications, HHT-genotype, and organ vascular malformations (VMs) will be measured. The data, aggregated as mean change from baseline using the scale, will enhance understanding and accelerate the development of new diagnostic and treatment options for HHT.

SECONDARY OUTCOMES:
Identify severe morbidity and mortality outcomes related to HHT using HHT Clinical Outcomes Scale | 10 years
  Description: Utilizing the "HHT Clinical Outcomes Scale," this measure aims to prospectively and longitudinally assess severe complications in HHT. This measure focuses on measuring rates of severe complications in HHT. Determinants of these complications will be characterized, and the data will be aggregated as mean change from baseline using the index, providing valuable insights into the disease progression.
Epistaxis Characterization with Epistaxis Severity Scale | 10 years
  Description: Utilizing the "Epistaxis Severity Scale," this measure aims to characterize epistaxis in adults with HHT, considering aspects such as frequency, duration, intensity, and variability. Outcome determinants related to epistaxis will be elucidated, and the data will be aggregated as mean change from baseline using the scale to inform comprehensive patient care.
Organ Vascular Malformation (VM) Development and Growth Assessment using Organ VMs Assessment Tool | 10 years
  Utilizing the "Organ VMs Assessment Tool," this measure involves the prospective measurement of the development and growth of organ vascular malformations (VMs) in HHT patients over time. Outcome determinants related to these VMs will be investigated, and the data will be aggregated as mean change from baseline using the tool, contributing to a better understanding of disease progression.
Treatment Outcomes Assessment with HHT Treatment Outcomes Scale | 10 years
  Utilizing the "HHT Treatment Outcomes Scale," this measure involves the prospective measurement of treatment outcomes for HHT and its clinical manifestations. Treatment outcome determinants will be characterized, and the data will be aggregated as mean change from baseline using the scale to guide effective management strategies for patients with HHT.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Dickey, MSN, Principal Investigator — Cure HHT
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Augusta University, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided